CLINICAL TRIAL: NCT06767189
Title: Preventing Recurrent Cardioembolic Stroke - Right Approach, Right Patient (The PRECISE Study)
Brief Title: Preventing Recurrent Cardioembolic Stroke (The PRECISE Study)
Acronym: PRECISE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Alan C Cameron, Dr, University of Glasgow
Other Study IDs: GN21ST183
Record Dates: First submitted 2025-01-06; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and buffy coat
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ECG monitoring — R-test or ECG patch for up to 28 days

SUMMARY:
Heart rhythm monitors are worn for 3 days after a stroke to look for an abnormal heart rhythm called atrial fibrillation (AF) that increases the risk of blood clots and second strokes. If AF is found, then blood thinning drugs called anticoagulants can greatly reduce the chance of a second stroke. However, there are often long waits for these tests to be done and only 4 out of every 100 people who have a 3 day heart rhythm monitor are found to have AF.

New heart rhythm monitors that are worn for longer find many more people with AF, but these tests are expensive and are not needed for all people after stroke. It has also been difficult to implement them in the NHS as a lot of time and resource is spent trying to perform 3 day heart rhythm monitors.

A solution is to identify people who are very unlikely to have AF after stroke and who do not need heart rhythm monitors for 3 days or longer. This will free resources to allow longer heart rhythm monitors to be focused on people who are more likely to have AF and benefit.

We aim to develop a risk score that highlights people who are unlikely to have AF after stroke, and who do not need heart rhythm monitors for 3 days or longer. We will use the risk score to develop a more personalised care pathway to look for AF after stroke that could reduce testing for many people after stroke. This would allow higher risk people to benefit from longer cardiac monitoring, increase AF detection rates and allow more people to benefit from anticoagulant drugs to prevent second strokes.

We will recruit 675 people admitted to hospital with a stroke who are not known to have AF. We will collect clinical information, heart rhythm recordings performed at rest (electrocardiograms/ECGs) and a blood to measure levels of the blood markers MRproANP, NTproBNP and genetic information. Everyone will have a 28 day heart rhythm monitor to search for AF.

We will analyse the clinical information, ECG recordings, MRproANP/NTproBNP levels and genetic data to develop a risk score that highlights people who do not have AF after 30 days of heart rhythm monitoring. We will use the risk score to develop a more personalised care pathway to search for AF after stroke that reduces the number of 3 day heart rhythm monitors performed and frees resources to focus longer heart rhythm monitoring on higher risk people who are more likely to benefit. We will assess the potential impact on healthcare costs of adopting this approach by estimating the number of second strokes that could be prevented by increased use of anticoagulant drugs for people who are found at have AF.

DETAILED DESCRIPTION:
Cardiac rhythm monitoring is performed to search for atrial fibrillation (AF) after ischaemic stroke or transient ischaemic attack (TIA). Prolonged cardiac rhythm monitoring increases AF detection but is challenging to implement in many healthcare settings and is not needed for all people after ischaemic stroke/TIA. We aimed to develop a model that includes clinical, electrocardiogram (ECG), blood-based, and genetic biomarkers to identify people with a low probability of AF detection after ischaemic stroke or TIA. We will recruit 675 consenting participants who are aged over 18 years, who were admitted with ischaemic stroke or TIA in the 5 days prior, who are not known to have AF, and who would be suitable for anticoagulation if AF is found. We will collect baseline demographic and clinical data, a 12-lead ECG, and a venous blood sample for blood biomarkers (including midregional pro-atrial natriuretic peptide, MRproANP; and N-terminal pro B-type natriuretic peptide, NTproBNP) and genetic data. We will perform up to 28 days of cardiac rhythm monitoring using an R-test or patch device to search for AF in all participants. The sample size of 675 participants is based on true sensitivity of 92.5%, null hypothesis sensitivity of 80%, 80% power, and 5% significance. The primary outcome is AF detection ≥30 s duration. Secondary outcomes are recurrent cardiovascular events and mortality. The results will guide the development of a more personalized care pathway to search for AF after ischaemic stroke or TIA. This could help to reduce cardiac rhythm monitoring for people with a low probability of AF detection and allow more intensive cardiac monitoring to be focused on people who are more likely to have AF and benefit. Participants will be consented for their data to be used in future research studies, providing a rich resource for stroke and cardiovascular research communities.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years Admitted with acute ischaemic stroke or TIA in the 5 days prior to enrolment No known AF Venous blood sampling possible Able to provide informed consent

Exclusion Criteria:

Contraindication to oral anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People admitted to hospital with acute ischaemic stroke or TIA who are not known to have AF and who would be suitable for treatment with anticoagulant drugs if AF is found.
Sampling Method: Non-Probability Sample
Enrollment: 675 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Atrial Fibrillation | 1 year
  AF Detection

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - NHS Lothian, Dundee
  - NHS Greater Glasgow and Clyde, Glasgow
  - NHS Lanarkshire, Glasgow